CLINICAL TRIAL: NCT06908187
Title: Parent Training for Autistic Toddlers: Development and Preliminary Testing
Brief Title: Opt-In Early Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Connecticut Children's Medical Center (Other); University of Connecticut (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Katharine Zuckerman, MD MPH, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00025956; R34MH132712 (NIH); no number (Other Grant/Funding Number: KUNI Foundation)
Record Dates: First submitted 2025-03-14; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Now - Latinx (Experimental): Families assigned to the Intervention Now group will receive the Opt-in Early online curriculum/website in their preferred language(s). Opt-in Early is a self-directed parent-training program targeting cognitive, language, social, and adaptive behaviors in children with new or suspected autism diagnoses. It is a mobile-device compatible website that can be accessed on any smart phone, tablet, or PC. The program is designed to bridge the time between when autism is first identified and when a child accesses more definitive services. It can also be used by parents who do not desire, or who cannot access in-person services. The program is publicly available and has 6 core modules and 6 optional modules, each of which takes ~1 hour to complete, as well as a detailed resource guide. It can be offered by primary care practices, autism specialty clinics, and educational programs, and requires minimal family support.
  Interventions: Other: Opt-In Early Latinx intervention
- Intervention Later (Control) (No Intervention): Families randomized to Intervention Later (control arm) will be offered (a) viewing of a 7-minute English or Spanish Youtube video about autism evaluation and treatment options (b) print educational materials (5th-grade reading level) about developmental delays, the meaning of screening positive for possible autism, and how to navigate the Early Intervention system in their state (Oregon or Connecticut), and (c) English or Spanish versions of the Autism Speaks First Concerns to Action Kit.
- Intervention Now - Rural (Experimental): Families assigned to the Intervention Now group will receive the Opt-in Early online curriculum/website in their preferred language(s). Opt-in Early is a self-directed parent-training program targeting cognitive, language, social, and adaptive behaviors in children with new or suspected autism diagnoses. It is a mobile-device compatible website that can be accessed on any smart phone, tablet, or PC. The program is designed to bridge the time between when autism is first identified and when a child accesses more definitive services. It can also be used by parents who do not desire, or who cannot access in-person services. The program is publicly available and has 6 core modules and 6 optional modules, each of which takes ~1 hour to complete, as well as a detailed resource guide. It can be offered by primary care practices, autism specialty clinics, and educational programs, and requires minimal family support.
  Interventions: Other: Opt-In Early Rural Intervention

INTERVENTIONS:
Other: Opt-In Early Latinx intervention — Participants will access to the Opt-In Early training program website, but will be able to access the Spanish language version as well. Families will fill out a usage diary to record their experience.
  Arms: Intervention Now - Latinx
Other: Opt-In Early Rural Intervention — Participants will access to the Opt-In Early training program website. Parents will be able to interact with the rural community-oriented aspects of the program. Families will fill out a usage diary to record their experience.
  Arms: Intervention Now - Rural

SUMMARY:
Latinx and Rural-living children with diagnosed or suspected autism have especially long wait times for diagnoses and intervention, up to a year or even more. This delayed access to intervention is likely to prevent children from reaching their full potential in skills and adaptive functioning. A comprehensive, online mobile device-based, free intervention that can be used by parents while on these wait lists may optimize their child's development. The investigators have developed such a program, the Online Parent Training in Early Intervention (OPT-In-Early) program. It teaches parents the fundamental principles of both applied behavior analysis and naturalistic interventions, uses non-technical language, video demonstrations, guidance in selecting appropriate skills to teach, embedding teaching into daily routines, and reducing interfering behaviors. It is a self-paced, individualized platform giving parents strategies to strengthen the parent-child relationship, to teach basic skills, such as simple communication, to reduce interfering behaviors, and to establish helpful routines. In pilot the RCT, parents (half of whom were self-identified as Latinx) rated the program very highly and showed positive changes in behavior and knowledge. The goal of the current project is to develop, and pilot test a bilingual Spanish/English culturally tailored version of OPT-In-Early for Latinx families in the US, as well as tailoring and testing the program for rural communities of Oregon. First, the investigators will obtain detailed, iterative feedback from bilingual Latinx parents with an autistic child regarding OPT-In-Early. Similar feedback will also be obtained from participants from rural communities of Oregon who also have an autistic child. The investigators will use this feedback to culturally adapt the program content and format. Next, the adapted program will be modified via user testing with Spanish speaking parents and English speaking parents. Finally, the bilingual version will be tested in a six-month pilot RCT, in preparation for a fully powered R01 trial. The investigators will use a wait-list control design: the Intervention Now arm will be given the online program and the Intervention Later arm (controls) will be given educational material about autism. All children will receive a baseline and 6-month follow-up assessment, which will measure parent fidelity in using the intervention principles (the primary outcome), child social communication, level of autism symptoms, impact of autism symptoms, and degree of developmental delays. The Intervention Now group will have two subgroups. One will test the online program with an emphasis placed on the Spanish version, while the other will focus on the English version and complete the program through a rural lens. At the conclusion of this research, the investigators will have developed an evidence-based, comprehensive, freely available, parent-delivered intervention that can be used by US Latinx and rural families on their mobile devices as they await diagnosis and intervention. This will increase parent efficacy and reduce their stress, accelerate children's skills, reduce interfering behavior, and enhance PCPs' willingness to implement universal autism screening.

ELIGIBILITY:
Inclusion Criteria:

* Parent-child dyads where the child has a definitive or provisional diagnosis of autism
* Children must be aged 15 - 42 months
* Latinx arm parents must be primarily Spanish-speaking or balanced bilinguals
* Rural arm participants would ideally reside in primarily rural communities (identified with RUCA codes; RUCA score >5)

Exclusion Criteria:

* Diagnosed with another major developmental condition (e.g., Down Syndrome, Hearing Impairment)

Min Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Social Interaction Rating Scale (SIRS) | It is administered pre- and post-six months of intervention to both groups.
  It is a measure of observed parent use of intervention strategies, to assess Parent Fidelity. This is observational measure is videotaped and coded by a trained rater blind to group. Parents are asked to do 4 activities with their child, keeping the child as engaged as possible: (1) Work on a puzzle (2) Teach your child to imitate you doing a simple behavior that you haven't already taught them to imitate; (3) Play with your child using bubbles. (4) Feed your child a snack. Each activity is recorded for 3 minutes. Parents' responsivity to the child based on behavioral and affective principles emphasized throughout OPT-In- Early are coded: positive affect, contingent reinforcement, appropriate directiveness, promotion of eye contact, and appropriate level of prompting. Each item is scored on a 5-point Likert scale Scores on the 5 items are also summed to yield a total score. OPT-In-Early pilot data demonstrated good-to-excellent ICC's for between-rater reliability for these SIRS items.

SECONDARY OUTCOMES:
Autism Impact Measure (AIM) | Once at baseline evaluation and a second at the end of the six months of intervention.
  It is a parent rating of core autism symptom. The AIM is one of few autism measures designed specifically to assess change in core symptoms due to treatment, and is sensitive to change over short-term treatment. For each symptom or developmental milestone listed, the parent indicates the frequency of the behavior and the impact that the parent thinks it has on the child's everyday functioning Western Psychological Services (the publisher) has already translated this instrument into Spanish. We are applying for permission to use this as a research instrument to WPS. . Improvement in child core autism symptoms will be assessed via changes in parent ratings of frequency and impact on functioning between the two administrations, the first at the baseline evaluation and the second at the end of the six months of intervention
Brief Observation of Social Communication Change (BOSCC) | It is administered at the baseline evaluation and after the six months of intervention or psycho-education.
  Change in child social communication is assessed via direct observation with the BOSCC, which detects subtle and short term changes in child social communication, unlike instruments that were primarily designed for diagnosis and may not be sensitive to short term or smaller changes (e.g., ADOS-2, BOSA, Tele-ASD-Peds). Furthermore, it can be administered by parents with RA instruction (not requiring a research reliable clinician) with a standard toy set. It is being used with guidance from the authors, in our just concluded NIH-funded ACE Connect the Dots study (Robins, PI, NICHD: 1R01MH115715); we are ready to have the RAs instruct the parents in the simple social presses and to bring a sanitized toy set to the assessment sessions. The authors have outlined procedures by which the very general parent instructions can be translated into parents' first language. BOSCC sessions, which are about 12 minutes long, are videotaped and coded by a trained RA blind to group.
Early Intervention Parenting Self-Efficacy Scale (EIPSES) | Responses are averaged across items to produce a single parenting self-efficacy score at the baseline evaluation and at the six month post-treatment evaluation.
  This a brief self-report measure of parents' perceptions of their parenting competence, and their ability to contribute to intervention outcomes for their children. The EIPSES has good internal consistency and adequate convergent validity (Guimond et al., 2008). A few Items were modified slightly by study investigators to be applicable to an intervention delivered to young children by caregivers. Senior author of the scale (Jeanne Wilcox, Prof. Emerita, ASU) gave us permission to translate the scale into Spanish.
Parenting Stress Index (PSI-4) | It is administered at the baseline evaluation and at the six month post-treatment evaluation.
  This index assesses parent stress; it is composed of 36 items, over 3 domains: Parental Distress, Parent Child Dysfunctional Interaction, and Difficult Child, which combine to form a Total Stress scale. The publisher has made the PSI available in Spanish.

OTHER OUTCOMES:
Treatment Evaluation Inventory - Short Form (TEI-SF) | It will be administered to parents in the intervention group after they have 6-month access to the material.
  This is a 9-item measure of acceptability of different aspects of treatment; it will be applied to each module, as in our prior pilot trial (Dai et al, 2021) for parents in the intervention group. Parents are instructed to rate any modules that they used. We previously translated this measure into Spanish with permission of the original first author, including addition of several items measuring cultural responsivity.
System Usability Scale (SUS) | Completed at the end of the intervention.
  The usability of the mobile platform will be assessed via the 10-item System Usability Scale (SUS) (Lewis, 2018), completed at the end of the intervention. This scale has been validated in Spanish and is widely used to assess usability of mobile applications and websites.
Intervention Uptake via Usage Diary | Multiple times throughout intervention.
  Parents will note date/time that they begin to view/read a specific module. Parents also enter an ID when they log on, and the program will track parents' opening each module, and requires re-log on after 30 minutes of non-use.
Initial Autism Severity measured via the Toddler Autism Symptom Inventory (TASI) | . It will be administered as part of the baseline evaluation and again after the six months of intervention.
  The TASI is a developmentally appropriate caregiver interview for use in diagnostic evaluations of toddlers that offers clearly operationalized diagnostic criteria, presence and absence of skills and autism symptoms, in children aged 12-36 months. Reliability and validity of items and a cutoff score for likelihood of autism spectrum disorder were established (Coulter et al, 2021a, 2024). Specificity and sensitivity of this cutoff were confirmed with a cross-validation sample. The TASI effectively identifies most children with DSM-5 autism with few false positives. The cut-off score will be used to determine threshold for probable autism, and the total score will serve as an estimate of autism severity.
Vineland Adaptive Behavior Scales, Third Edition: Survey Interview Form | Administered six months after receiving intervention.
  The Vineland-3 is a standardized, well-used, parent interview designed to measure adaptive behaviors in the domains of Communication, Daily Living Skills, Socialization, and Motor Skills. Internal consistency is excellent and inter-rater reliability is good (Sparrow et al., 2016). Standard scores in Communication and Socialization domains are used to quantify children's baseline adaptive functioning in both groups. The Vineland is available in Spanish. Six months after the intervention group parents are given access to the parent training program, and the control group parents are given the psycho-educational materials, the Vineland will be re-administered by a trained RA blind to group. Change scores for each child will be the difference in standard scores on Communication and Socialization.
Opt-In-Early Knowledge Check | Completed at baseline and immediately after the intervention.
  The study investigators created a multiple choice quiz to assess knowledge of the content covered in the first six (mandatory) modules of OPT-In-Early. The quiz was created without using the module content verbatim and therefore required the ability to understand and apply the principles taught.
Child and Family Demographics | Obtained by survey on enrollment.
  Demographics will be obtained by survey on enrollment, including caregiver age, gender, race, education, and child age, sex, and ethnicity, as well as insurance type and other autism services being received. These items will be adapted from the U.S. Census American Community Survey and the National Survey of Children's Health. All items have been validated in Spanish. English proficiency, national origin and Spanish language dominance will be measured through the Bilingual Language Profile.
Initial Concern adapted from the ADI-R | All participants will receive these measures at the beginning of the study.
  Three questions about first concerns were adapted from the ADI-R (Herlihy et al, 2015): age of first concern, nature of concern (with a list of ASD-specific and non-ASD-specific concerns), and magnitude of concern (on a Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Zuckerman, MD MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided
We will be submitting data to NIMH NDA archive as required by the funder

REFERENCES:
- [Background] Ruble, L., McDuffie, A., King, A. S., & Lorenz, D. (2008). Caregiver responsiveness and social interaction behaviors of young children with autism. Topics in Early Childhood Special Education, 28(3), 158-170
- [Background] Nielsen J. Usability Engineering. San Diego, CA: Academic Press; 1993.
- [Background] Mazurek MO, Carlson C, Baker-Ericzen M, Butter E, Norris M, Kanne S. Construct Validity of the Autism Impact Measure (AIM). J Autism Dev Disord. 2020 Jul;50(7):2307-2319. doi: 10.1007/s10803-018-3462-8. PMID 29344761
- [Background] Mazurek MO, Carlson C, Baker-Ericzen M, Butter E, Norris M, Barr C, Kanne S. The Autism Impact Measure (AIM): Examination of Sensitivity to Change. Autism Res. 2020 Nov;13(11):1867-1879. doi: 10.1002/aur.2397. Epub 2020 Oct 1. PMID 33001561
- [Background] Kelley, M. L., Hefer, R. W., Gresham, F. M., & Elliott, S. N. (1989). Development of a modified treatment evaluation inventory. Journal of Psychopathology and Behavioral Assessment, 11(3), 235-247.
- [Background] Kanne SM, Mazurek MO, Sikora D, Bellando J, Branum-Martin L, Handen B, Katz T, Freedman B, Powell MP, Warren Z. The Autism Impact Measure (AIM): initial development of a new tool for treatment outcome measurement. J Autism Dev Disord. 2014 Jan;44(1):168-79. doi: 10.1007/s10803-013-1862-3. PMID 23748386
- [Background] Herlihy L, Knoch K, Vibert B, Fein D. Parents' first concerns about toddlers with autism spectrum disorder: effect of sibling status. Autism. 2015 Jan;19(1):20-8. doi: 10.1177/1362361313509731. Epub 2013 Nov 11. PMID 24216070
- [Background] Guimond, A. B., Wilcox, M. J., & Lamorey, S. G. (2008). The Early Intervention Parenting SelfEfficacy Scale (EIPSES) scale construction and initial psychometric evidence. Journal of Early Intervention, 30(4), 295-320
- [Background] Grzadzinski R, Lord C. Commentary: Insights into the Development of the Brief Observation of Social Communication Change (BOSCC). J Ment Health Clin Psychol. 2018;2(5):15-18. doi: 10.29245/2578-2959/2018/5.1166. Epub 2018 Oct 9. No abstract available. PMID 30854524
- [Background] Grzadzinski R, Carr T, Colombi C, McGuire K, Dufek S, Pickles A, Lord C. Measuring Changes in Social Communication Behaviors: Preliminary Development of the Brief Observation of Social Communication Change (BOSCC). J Autism Dev Disord. 2016 Jul;46(7):2464-79. doi: 10.1007/s10803-016-2782-9. PMID 27062034
- [Background] Dai YG, Thomas RP, Brennan L, Luu ML, Hughes-Lika J, Reilly M, Moreno P, Obe B, Ahmed KB, Berry LN, Goin-Kochel RP, Helt MS, Barton ML, Dumont-Mathieu T, Robins DL, Fein DA. An initial trial of OPT-In-Early: An online training program for caregivers of autistic children. Autism. 2023 Aug;27(6):1601-1615. doi: 10.1177/13623613221142408. Epub 2022 Dec 15. PMID 36519775
- [Background] Dai YG, Thomas RP, Brennan L, Helt MS, Barton ML, Dumont-Mathieu T, Fein DA. Development and Acceptability of a New Program for Caregivers of Children with Autism Spectrum Disorder: Online Parent Training in Early Behavioral Intervention. J Autism Dev Disord. 2021 Nov;51(11):4166-4185. doi: 10.1007/s10803-020-04863-z. Epub 2021 Feb 2. PMID 33527164
- [Background] Dai YG, Brennan L, Como A, Hughes-Lika J, Dumont-Mathieu T, Rathwell IC, Minxhozi O, Aliaj B, Fein DA. A Video Parent-Training Program for Families of Children with Autism Spectrum Disorder in Albania. Res Autism Spectr Disord. 2018 Dec;56:36-49. doi: 10.1016/j.rasd.2018.08.008. Epub 2018 Sep 10. PMID 31275428
- [Background] Birdsong, D., Gertken, L. M., & Amengual, M. (2012). Bilingual language profile: An easy-to-use instrument to assess bilingualism. COERLL, University of Texas at Austin.
- [Background] Abidin, R. (2012). Parenting Stress Index™, Fourth Edition Short Form. Lutz, Florida: Psychological Assessment Resources.